CLINICAL TRIAL: NCT03917771
Title: Study to Evaluate the Efficacy of Early Detection of Lower Extremity Lymphedema After Lymphadenectomy in Gynecological Cancer and Implantation of the Protocol
Brief Title: Early Detection of Lower Extremity Lymphedema After Lymphadenectomy in Gynecological Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Donostia (Other)
Responsible Party: Principal Investigator, IBON JAUNARENA, Oncology Gynecologist, Hospital Donostia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IJM-EDL- 2017-01
Record Dates: First submitted 2018-08-16; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Lymphedema of Limb; Sentinel Lymph Node
Keywords: physiotherapy

STUDY DESIGN:
Intervention Model Description: Recruitment Process: patients will be selected consecutively and offered to participate in the study
Who Masked: Outcomes Assessor
Masking Description: randomization according to system of envelopes with code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early lymphedema detection (Experimental): Face-to-face consultation in Rehabilitation for early detection of lymphedema after surgery. Lower Limb measurement and care education
  Interventions: Other: Early lymphedema detection
- Usual follow-up (Active Comparator): The usual follow-up will be carried out in GO consultation (0,1,6,12 months)
  Interventions: Other: Usual follow-up

INTERVENTIONS:
Other: Early lymphedema detection — Face-to-face consultation in Rehabilitation for early detection of lymphedema after surgery (1,6,12 months). Lower Limb measurement and care education
  Arms: Early lymphedema detection
Other: Usual follow-up — Usual follow-up carried out in GO consultation
  Arms: Usual follow-up

SUMMARY:
This study aims to detect and treat early lower limb lymphedema secondary to lymphadenectomy with the aim of increasing the quality of life of patients with this chronic condition.

To this end, a group of patients (treatment group) will be referred to the Rehabilitation service for a previous consultation and after surgery where lymphedema could be detected early. In addition, the usual follow-up will be carried out in Gynecology Oncology consultation (GO). In the second group, also called control, will be performed the usual follow-up in GO.

For this we randomize to one of these two groups. The research project has the favorable report of the Center's Clinical Research Ethics Committee

DETAILED DESCRIPTION:
METHODOLOGY:

1. Type of study: A) Randomized clinical trial B) Prospective cohort observational study
2. Study period: from January 2017 to December 2017.
3. Scope: health area of the province of Gipuzkoa and the University Hospital of Donostia as a reference center.
4. Selection of the population:

   4.1. The inclusion criteria will be: A) Diagnostic gynecological cancer patients submitted to bilateral laparoscopic pelvic lymphadenectomy as laparotomics (B: Sentinel Node Biopsy study, SNB) within the usual surgical protocol, with expected survival greater than 12 weeks and adequate liver, renal and medullary functions to accept And sign informed consent 4.2. The exclusion criteria for the study will be: Blood clotting or hematological disorders, previous thromboembolic disease and history of lymphatic system disease (lymphedema or lymphocele), contraindication for physiotherapy or who do not wish to participate and / or do not sign informed consent.

   4.3. Sample size: A) Assuming that according to previous studies the overall incidence of lymphedema after LPL is 21% (Hareyama et al), its estimated that a minimum sample of 44 patients will bi needed in order to be able to demonstrate at least 4-fold detection (Torres et al) of Lymphedemas with early follow-up with alpha = 0.05 and beta = 0.2, estimating that habitual follow-up detects 13% of lymphedema ( Mohler III et al).

   4.4. Recruitment Process: Will be selected consecutively and offered to participate in the study.
5. 5.1 Intervention: A) After diagnosis and programming for surgery at the GO consultation, circometry is performed by a trained nurse. During the admission, the nurse delivers and explains recommendations sheet and is offered to participate in the clinical trial giving him the Informed Consent (IC) and Information Sheet created for this purpose. In case of accepting and signing the IC, it is randomized (total randomization) according to system of envelopes with code.

Distribution of the intervention;

* Treatment group: Face-to-face consultation in Rehabilitation for early detection of lymphedema after surgery (1,6,12 months). Lower Limb measurement and care education
* Control group: The usual follow-up will be carried out in GO consultation (0,1,6,12 months)

The pelvic lymphadenectomy will be performed by the same surgical team using a transperitoneal approach. The limits of lymph node dissection will be: the psoas muscle, laterally, the postero-medially internal iliac artery, the bifurcation of the common iliac artery cranially, where it crosses the ureter, and caudally the origin of the epigastric vessels, to level of the deep circumflex iliac vein.

B) After diagnosis and programming for surgery at the GO consultation, circometry is performed by trained and yearly nurse. During the entrance, it is delivered and explains the recommendations sheet. SNB is performed by detecting sentinel ganglion from the above mentioned areas according to the protocol of the service. The usual follow-up will be carried out in GO consultation (0,1,6,12 months)

ELIGIBILITY:
Inclusion Criteria:

* A) Diagnostic gynecological cancer patients submitted to bilateral laparoscopic pelvic lymphadenectomy as laparotomics (B: Sentinel Node Biopsy study, SNB) within the usual surgical protocol, with expected survival greater than 12 weeks and adequate liver, renal and medullary functions to accept And sign informed consent

Exclusion Criteria:

* The exclusion criteria for the study will be: Blood clotting or hematological disorders, previous thromboembolic disease and history of lymphatic system disease (lymphedema or lymphocele), contraindication for physiotherapy or who do not wish to participate and / or do not sign informed consent.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of the implantation of a standardized postoperative follow-up for the early detection of lymphedema secondary to lymphadenectomy in gynecological cancer | 12 months
  Lower Limb measurement secondary to lymphadenectomy in gynecological cancer

SECONDARY OUTCOMES:
Implementation of educational strategy for patients and professionals | 12 months
  Care education questionnaire results

CONTACTS AND LOCATIONS:
Overall Officials: IBON JAUNARENA, Principal Investigator — Hospital Donostia
Locations (1):
- Donostia Hospital, San Sebastián, Gipuzkoa, Spain